CLINICAL TRIAL: NCT03841916
Title: The Relationship Between Transvaginal Ultrasound Endometrial Thickness and Body Mass Index and Pathology in Postmenopausal Bleeding
Brief Title: Relation Between Body Mass Index and Endometrial Thickness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Kasr El Aini Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Body mass index
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Postmenopausal Bleeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: transvaginal ultrasound — transvaginal ultrasound to measure endometrial thickness

SUMMARY:
Postmenopausal Bleeding (PMB) is defined as recurrent attacks of bleeding occurring in women after menopause one year at least after stoppage of cycles [

DETAILED DESCRIPTION:
Premalignant lesions and malignant lesions most commonly complex hyperplasia with atypia and carcinoma of the endometrium are present in 1/3 of patients evaluated for postmenopausal bleed-ing, and so investigations for cases of postmeno-pausal bleeding are mandatory

ELIGIBILITY:
Inclusion Criteria:

* menopausal women (defined as minimum of 1 year of amenorrhea after the age of 45 years if only the amenorrhea is not related to pregnancy, medication or disease),

Exclusion Criteria:

* Women with chronic diseases as diabetes mellitus, hypertension or hematological disorders, those received hormone replacement therapy, Tamoxifen or anticoagulant therapy and women with adnexal massed detected by TVUS or apparent causes of bleeding from cervix or vagina e.g. ulcer were excluded.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — women who have postmenopausal bleeding
Study Population: women with postmenopausal bleeding
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-12-02 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-03-20 (Estimated)

PRIMARY OUTCOMES:
the number of women who will have a relation between endometrial thickness and BMI | within 2 weeks
  if there is a relation between increased BMI and endometrial thickness

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, PhD, Principal Investigator — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt
Locations (1):
- Algazeerah and Kasralainy hospital, Giza, Egypt